CLINICAL TRIAL: NCT02391051
Title: Focal Brachytherapy in Patients With Selected "Low-risk" Prostate Cancer - a Phase-II-trial
Acronym: FOKAL-BT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOKAL-BT
Record Dates: First submitted 2014-07-01; First posted 2015-03-18 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; focal brachytherapy; PSA; Biological marker
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Focal Brachytherapy (Experimental): HDR-Brachytherapy, 2 fractions within at least 24 but max. 30 hours, each 13,5 Gy
  Interventions: Radiation: HDR-Brachytherapy

INTERVENTIONS:
Radiation: HDR-Brachytherapy — HDR-Brachytherapy 2x 13,5 Gy

SUMMARY:
This trial examines the feasibility and toxicity of focal brachytherapy in patients with low-risk prostate cancer.

DETAILED DESCRIPTION:
Patients with low-risk prostate cancer will receive HDR-Brachytherapy: 2 x 13,5 Gy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Histologically confirmed prostate cancer
* Gleason Score of index lesion ≤ 6 (3+3)
* Tumor stage: cT1-2a cN0 cM0
* Unilateral affection; index lesion ≤ 0.5ml with or without clinically non-significant lesion contralateral. No more than 25% of the punch should be affected. Therefore a 3D-TPM-biopsy is mandatory before treatment.
* PSA ≤ 10/ng/ml
* Prostate volume < 60 m^3
* No distant metastasis
* Life expectancy > 10 years
* Informed consent

Exclusion Criteria:

* Tumor stage ≥ T2b
* Known metastasis: N+ and/or M1
* General anesthesia or peridural anesthesia is not possible
* Coagulation disorder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-10; Primary Completion 2019-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Intensity and frequency of adverse events | 6 weeks after therapy

SECONDARY OUTCOMES:
Tumor regression | 6 weeks up to 10 years after therapy
Rate of recurrences measured by PSA | 10 years after therapy
Correlation of Markers RTEN, ERG, APN, Ki67, KPNA1, PSMA, FGFR1, PMP22, CDKN1A/P16, PDCD4, KLF6, PITX with PSA free survival | 10 years after therapy
Correlation of microRNA141 and -375 with outcome | 10 years after therapy
Feasibility, as measured by NCI-CTCAE-scale, EORTC-QLQ, IIEF, IPSS, ICIQ | 6 weeks after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Vratislav Strnad, MD, Study Chair — University Hospital Erlangen, Dept. of Radiooncology; Bastian Keck, MD, Study Chair — University Hospital Erlangen, Dept. of Urology; Alexander Cavallaro, MD, Study Chair — University Hospital Erlangen, Dept. of Radiology; Arndt Hartmann, MD, Study Chair — University Hospital Erlangen, Dept. of Pathology; Michael Lotter, Dipl.-Phys., Study Chair — University Hospital Erlangen, Dept. of Radiooncology; Annedore Strnad, MD, MHBA, Study Chair — University Hospital Erlangen, Dept. of Radiooncology; Peter Goebell, MD, Study Chair — University Hospital Erlangen, Dept. of Urology; Wolfgang Uter, MD, Study Chair — University Erlangen; Dept. of Biometrics and Epidemiology; Michael Uder, MD, Study Chair — University Hospital Erlangen, Dept. of Radiology; Bernd Wullich, MD, Study Chair — University Hospital Erlangen, Dept. of Urology; Rainer Fietkau, MD, Study Chair — University Hospital Erlangen, Dept. of Radiooncology
Locations (1):
- University Hospital, Erlangen, Germany